CLINICAL TRIAL: NCT03259984
Title: Epigenetics and the Origin of Muscle Insulin Resistance in Humans Aims 1-3
Brief Title: Epigenetics of Muscle Insulin Resistance
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Dawn K Coletta, Associate Professor of Medicine, University of Arizona
Other Study IDs: 1612045470
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from vastus lateralis skeletal muscle biopsies and blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1: This experiment will use the next generation sequencing reduced representation bisulfite sequencing to define patterns of DNA methylation in skeletal muscle and whole blood tissue of metabolically well-characterized lean healthy, obese nondiabetic, and type 2 diabetic volunteers. The investigators will test the hypotheses that: (a) There is an increased methylation of genes involved in mitochondrial biogenesis and oxidative phosphorylation and altered methylation of promoters of genes coding for extracellular matrix and cytoskeletal proteins in insulin resistance, (b) The altered methylation patterns observed correspond to protein and mRNA expression changes, and (c) There are coordinated patterns of DNA methylation between the skeletal muscle and whole blood tissues in insulin resistance.
- Aim 2: This experiment will test the hypotheses in lean healthy, obese non-diabetic and type 2 diabetic volunteers that: (a) Increased methylation of the PGC-1α promoter predicts a decreased response of this gene to a single bout of exercise, and (b) Altered methylation of promoters of nuclear encoded mitochondrial genes predicts a decreased response of this gene to a single bout of exercise.
- Aim 3: This experiment will test the hypothesis in lean healthy, obese non-diabetic and type 2 diabetic volunteers that: (a) There is decreased methylation of genes involved in mitochondrial biogenesis and oxidative phosphorylation, and the altered methylation corresponds to protein and mRNA (messenger ribonucleic acid) expression changes, (b) There is altered methylation of genes involved in inflammation and cytoskeletal structure.

SUMMARY:
The investigators are trying to understand the role of DNA (deoxyribonucleic acid) methylation in insulin resistance in skeletal muscle and blood tissues. DNA methylation is a normal chemical process in the body that modifies DNA. By studying this, the investigators hope to better understand the causes of insulin resistance.

DETAILED DESCRIPTION:
Insulin resistance is defined as the decreased ability of insulin to perform its biological function in the muscle, liver and fat. Genetic and environmental factors are known to influence insulin sensitivity. It is not known how this is mediated. This study looks at the role of epigenetics (modifications of proteins associated with DNA and methylation of DNA) in alterations in insulin resistance. The investigators will study lean healthy people, obese non-diabetic people and people with type 2 diabetes to characterize the DNA methylation patterns in muscle in each group. The second aim of the study is to see how a single bout of exercise affects the DNA methylation in the muscle. The third aim looks at the effect of 8 weeks of supervised exercise on the DNA methylation.

ELIGIBILITY:
Inclusion Criteria

1. Age 21-55
2. BMI: Lean, BMI less than or equal to 25; Obese, BMI between 30- 50; type 2 diabetic, BMI between 30- 50.
3. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
4. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
5. Subjects must range in age as described in each specific protocol.
6. Subjects must have the following laboratory values:

   1. Hematocrit ≥ 35 vol%
   2. Serum creatinine ≤ 1.6 mg/dl
   3. AST (SGOT) < 2 times upper limit of normal
   4. ALT (SGPT) < 2 times upper limit of normal
   5. Alkaline phosphatase < 2 times upper limit of normal
   6. Triglycerides < 150 mg/dl for nondiabetics
   7. Triglycerides <300 for diabetics
   8. INR ≤ 1.3

Exclusion Criteria

1. Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded. Patients with type 2 diabetes will be excluded if they are taking thiazolidinediones, but may be taking sulfonylureas or other medications known to work through effects on insulin secretion.
2. Subjects receiving Gemfibrozil must not also be receiving a statin.
3. Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
4. Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three groups of volunteers will be studied: 1) lean, healthy volunteers, 2) obese volunteers without type 2 diabetes, and 3) volunteers with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
DNA methylation of genes in insulin resistance | 9 months
  DNA methylation of genes involved in mitochondrial biogenesis, oxidative phosphorylation, extracellular matrix and cytoskeleton proteins in insulin resistance, with an acute episode of exercise, and with eight weeks of training exercise.

SECONDARY OUTCOMES:
mRNA expression of genes | 9 months
  mRNA expression of genes involved in mitochondrial biogenesis, oxidative phosphorylation, extracellular matrix and cytoskeletal signaling are altered in insulin resistance, with an acute episode of exercise and with 8 weeks of exercise training.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Coletta, Ph.D., Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No